CLINICAL TRIAL: NCT06503237
Title: Safety and Efficacy of SWK002 in Patients With D2T-Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SWKCART23071101
Record Dates: First submitted 2024-07-07; First posted 2024-07-16 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD19 CART (Experimental): Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CART infusion. A dose of Anti-CD19 CART will be infused on day 0.
  Interventions: Drug: Anti-CD19 CART cells will be given IV at split doses.

INTERVENTIONS:
Drug: Anti-CD19 CART cells will be given IV at split doses. — Split intravenous infusion of Anti-CD19 CART cells of (Dose escalating infusion of 1 - 6 x10^6 CART cells/kg).

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with refractory rheumatoid arthritis. This study aims to evaluate the safety and efficacy of the treatment with Anti-CD19 CART.

ELIGIBILITY:
Inclusion Criteria:

1. no gender restriction and age of 18 years and above at the time of signing the informed consent form.
2. written informed consent approved by the Ethics Committee must be signed in person by all subjects or guardians prior to the commencement of any screening procedure.
3. adult refractory patients who meet the 2010 ACR / EULAR RA diagnostic criteria, with refractory defined as (1) failure of treatment with csDMARDs (2) experiencing failure of treatment with ≥2 bDMARDs/tsDMARDs with different mechanisms of action (3) meeting one of the following criteria: 1) DAS28-ESR >3.2 or CDAI >10 2) inability to hormone Hormone cannot be reduced to less than 7.5mg/day (3) Number of swollen joints and/or painful joints ≥3.
4. Stable treatment with 1 or 2 cs DMARD ( s ) prior to enrollment as follows: (1) at least 12 weeks of methotrexate and at least 4 weeks of administration at a dose of 7.5-25 mg/week (2) at least 4 weeks of stable hydroxychloroquine dose of ≤400 mg/d (3) at least 4 weeks of stable oral salicylsulphadiazepine 1-3 g/d (4) at least 4 weeks of stable oral leflunomide 10-20 mg/day Methylphenidate 10-20 mg/d.
5. no active or latent tuberculosis.
6. Adequate organ function: (1) blood creatinine ≤1.5 times the upper limit of normal, or glomerular filtration rate (eGFR) ≥60m/min/1.73m2 as estimated by the MDRD formula (2) and ALT ≤ 5 times the upper limit of normal for the corresponding age and total bilirubin ≤ 2.0 mg/dl (3) and ≤ 1 grade of dyspnea and oxygen saturation > 91% in room air.
7. hemodynamically stable with a left ventricular ejection fraction (LVEF) ≥45% as determined by echocardiography or multichannel radionuclide angiography (MUGA).
8. female subjects of childbearing potential and all male subjects must agree to use a highly effective method of contraception until at least 12 months after SWK002 infusion and until two consecutive PCR assays show no more CAR-T cells in the body.

Exclusion Criteria:

1. malignant tumors.
2. subjects with current or history of CNS disorders such as seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
3. previous subjects who have undergone allogeneic hematopoietic stem cell transplantation (HSCT).
4. subjects who have received chemotherapy other than pretreatment chemotherapy within 2 weeks prior to infusion.
5. subjects who have received other investigational drug therapy within 30 days prior to signing the informed consent.
6. active hepatitis B (defined as hepatitis B surface antigen positivity or hepatitis B core antibody positivity combined with a hepatitis B virus DNA test value >1000 copies/ml) or hepatitis C (HCV RNA positivity) subjects.
7. HIV antibody positive or syphilis spirochete antibody positive subjects.
8. subjects with uncontrolled acute life-threatening bacterial, viral or fungal infections (e.g., positive blood cultures ≤ 72 hours prior to infusion).
9. subjects who have lost or donated more than 400 mL of blood within 2 months prior to screening or have received a blood transfusion.
10. any history of definite drug or food allergy, especially to drugs related to the therapeutic agents (e.g., fludarabine, cyclophosphamide) or product components (e.g., DMSO) used in this trial.
11. any systemic cytotoxic or systemic immunosuppressive agent within 6 months prior to screening or during the study period, or any localized cytotoxic or localized immunosuppressive agent within 30 days or 5 half-lives (whichever is longer) prior to screening or during the study period.
12. pregnancy (as determined by blood pregnancy test) or lactation.
13. prevalence of systemic inflammatory diseases other than RA (except secondary Sjogren's syndrome), including but not limited to juvenile chronic arthritis, Crohn's disease, ulcerative colitis, psoriatic arthritis, systemic lupus erythematosus, ankylosing spondylitis, reactive arthropathy, systemic vasculitis, or gout.
14. the existence of unstable angina pectoris and/or myocardial infarction in the 6 months prior to signing the informed consent.
15. other conditions that, in the opinion of the investigator, should not be enrolled in this clinical study, such as poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome | up to 2 years
  All adverse events (AEs) will be listed and summarized. Summaries of laboratory data will include, at a minimum, treatment-emergent laboratory abnormalities. Summaries of AEs and laboratory abnormalities will be based on the All Treated analysis set.

SECONDARY OUTCOMES:
The persistence, accumulation, and migration of Anti-CD19 CART cells | Day-1, 1, 3, 5, 7, 9, 11, 14, 21, 28 and Month 2, 3, 6, 9, 12
  Assessing the trafficking of Anti-CD19 CART cells in the peripheral blood at the time of each infusion as well as at each time of follow-up by Quantitative Real-time Polymerase Chain Reaction or flow cytometry. Peripheral blood will be collected prior to the initial infusion and will be set as baseline.
Erythrocyte Sedimentation Rate | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12
  To evaluate RA disease activity
American College of Rheumatology (ACR) criteria 20, 50, 70 response rate | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12
  To evaluate RA disease activity
Swollen and tender joint count | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12
  To evaluate RA disease activity
Visual Analogue Scale | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12
  The visual analogue scale is used to assess pain. The basic method is to use a swimming scale about 10cm long, marked with 10 scales on one side, and the two ends are "0" and "10" respectively, 0 points represent no pain, and 10 points represent the most unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Siweikang Therapeutic Co.Ltd, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No